CLINICAL TRIAL: NCT07312136
Title: Evaluating the Prevalence and Severity of MASLD in Primary Care - a Follow-up Study
Brief Title: MASLD in Type 2 Diabetes in Primary Care - a Follow-up Study
Acronym: EPSOMIP2
Status: Enrolling by invitation | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: University Hospital, Linkoeping (Other); Amra Medical AB (Industry)
Responsible Party: Principal Investigator, Patrik Nasr, Adj Associate Professor, Docent, Specialist doctor, Linkoeping University
Other Study IDs: 2024-05471-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Cirrhosis; Advanced Fibrosis; Sarcopenia; Obesity & Overweight; Type 2 Diabetes; Hypertension; OSAS (Obstructive Sleep Apneas Syndrome); Metabolic Syndrome
Keywords: MASLD; Fibroscan; PDFF; MRE; Obesity
MeSH Terms: conditions — Fibrosis; Sarcopenia; Obesity; Overweight; Diabetes Mellitus, Type 2; Hypertension; Sleep Apnea, Obstructive; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA, RNA, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The EPSOMIP2 (Evaluating the Prevalence and Severity Of MASLD In Primary care - a Follow-up Study) trial is a longitudinal cohort study of patients with type 2 diabetes recruited from primary health care centers in Östergötland, Sweden. Between 2019-2023, 317 patients were included and underwent rigorous clinical evaluation, vibration controlled transient elastography, biobanking of bloodsamples, and the latest magnetic resonance techniques to liver and body composition. All patients alive will be re-invited to undergo the same evaluation and additional tests.

ELIGIBILITY:
Inclusion Criteria:

* Previously included and fulfilled evaluation in EPSONIP trial (NCT03864510)
* Age >/= 18 years
* Informed consent

Exclusion Criteria:

* Contraindication to magnetic resonance
* Other primary liver disease than MASLD diagnosed after inclusion EPSONIP trial (NCT03864510)
* Liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who where previously included, and fulfilled participation, in the EPSONIP trial (NCT03864510) between 2019 and 2023 are re-invited to fulfill the same evaluation with additional tests.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of MASLD | 2031
  Number of patients with MASLD measured with MRI-PDFF or CAP
Progression/regression of MASLD | 2031
  Number of patients who progress/regress to/from MASLD between two timepoints as measured with MRI-PDFF or CAP
Predictors of MASLD progression/regression | 2031
  Liver fat measured with MRI-PDFF. Predicitive variables collected through clinical evaluation, blood tests, physical activitiy evaluation, OSAS evaluation, hypertension measurements among others.
Prevalence of advanced fibrosis | 2031
  Number of patients with advanced liver disease as defined by VCTE or MRE (or clinically, i.e., signos of cirrohsis or hepatic decompensation)
Progression/regression of advanced fibrosis | 2031
  Progression/regression to/from advanced liver disease as measured with VCTE or MRE between two timepoints
Predictors of fibrosis progression/regression | 2031
  Liver fibrosis measured with MRE or VCTE. Predicitive variables collected through clinical evaluation, blood tests, physical activitiy evaluation, OSAS evaluation, hypertension measurements among others.
The association between physical activity and prevalent advanced fibrosis | 2031
  Liver fibrosis measured with VCTE or MRE. Physical activity measured with the international fitness scale (IFIS) and/or Actigraph GT3X (accelerometer).
The association between physical activity and risk of progressing to advanced fibrosis | 2031
  Liver fibrosis measured with MRE or VCTE. Physical activity measured with the international fitness scale (IFIS) and/or Actigraph GT3X (accelerometer).
Genetic factors associated with advanced fibrosis or MASLD progression/regression | 2031
  Liver fibrosis measured with MRE and VCTE. Liver fat measured with MRI-PDFF and CAP. Genes to be analyzed: PNPLA3, TM6SF2, MBOAT among others.
Association between body composition and MASLD and/or liver fibrosis and progression/regression thereof | 2031
  Liver fat measured with MRI-PDFF or CAP. Liver fibrosis measured with MRE or VCTE. Body composition measured with AMRA Medical AB's MAsS Scan.

SECONDARY OUTCOMES:
The association of hypertension and MASLD (with or withour signs of advanced fibrosis) | 2031
  Liver fibrosis measured with MRE or VCTE. Hypertension measured with weekly blood pressure measurement and/or 24 hour blood pressure measurement.
The association between OSAS and MASLD (with or withour advanced fibrosis) | 2031
  Liver fat measured with MRI-PDFF or CAP. Liver fibrosis measured with VCTE or MRE. OSAS measured at university hospital sleep apnea.
Health economic model for disease management | 2034
  Markov modelling
Number of patients that develop symptoms of end-stage liver disease | 2035
  Symptoms of end-stage liver disease (ascites, encepahopathy, varices, HCC) or liver related Death will be recorded through chart review

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Nasr, M.D., Ph.D., Principal Investigator — Department of Health, Medicine and Caring Sciences, Linköping University, and Department of Gastroenterology and Hepatology, Linköping University Hospital, Linköping, Sweden
Locations (1):
- Department of Gastroenterology and Hepatology, Linköping University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided